CLINICAL TRIAL: NCT03840902
Title: A Multicenter, Double Blind, Randomized, Controlled Study of M7824 With Concurrent Chemoradiation Followed by M7824 Versus Concurrent Chemoradiation Plus Placebo Followed by Durvalumab in Participants With Unresectable Stage III Non-small Cell Lung Cancer
Brief Title: M7824 With cCRT in Unresectable Stage III Non-small Cell Lung Cancer (NSCLC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Based on recommendations by an external Independent data Monitoring Committee (IDMC), Sponsor decided to discontinue this clinical study due to a low likelihood of achieving superiority in the efficacy endpoints versus standard of care.
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MS200647_0005; 2018-003265-34 (EudraCT Number)
Record Dates: First submitted 2019-02-12; First posted 2019-02-15 (Actual); Results first posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small Cell Lung Cancer; Bintrafusp alfa (proposed INN); M7824; Durvalumab; Stage III; INTR@PID LUNG 005
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab; Etoposide; Pemetrexed; Carboplatin; Paclitaxel; Cisplatin; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- cCRT plus M7824 followed by M7824 (Experimental): Participants received cCRT: Cisplatin/Etoposide or Carboplatin/Paclitaxel or Cisplatin/Pemetrexed concomitant with Intensity Modulated Radiation Therapy (IMRT) along with M7824 followed by M7824.
  Interventions: Drug: M7824; Drug: Etoposide; Drug: Pemetrexed; Drug: Carboplatin; Drug: Paclitaxel; Drug: Cisplatin; Radiation: Intensity Modulated Radiation Therapy (IMRT)
- cCRT plus placebo followed by durvalumab (Active Comparator): Participants received cCRT: Cisplatin/Etoposide or Carboplatin/Paclitaxel or Cisplatin/Pemetrexed concomitant with Intensity Modulated Radiation Therapy (IMRT) along with placebo matched to M7824 followed by durvalumab.
  Interventions: Drug: Placebo; Drug: Durvalumab; Drug: Etoposide; Drug: Pemetrexed; Drug: Carboplatin; Drug: Paclitaxel; Drug: Cisplatin; Radiation: Intensity Modulated Radiation Therapy (IMRT)

INTERVENTIONS:
Drug: M7824 — Participants received intravenous infusion of 1200 milligram (mg) M7824 over 1 hour every 2 weeks (q2w) during cCRT and up to 1 year after cCRT until unacceptable toxicity, confirmed disease progression assessed by investigator.
  Arms: cCRT plus M7824 followed by M7824
Drug: Placebo — Participants received intravenous infusion of placebo matched to M7824 over 1 hour q2w during cCRT until unacceptable toxicity, confirmed disease progression assessed by investigator.
  Arms: cCRT plus placebo followed by durvalumab
Drug: Durvalumab — Participants received intravenous infusion of durvalumab 10 milligram per kilogram (mg/Kg) over 1 hour q2w up to 1 year after cCRT until unacceptable toxicity, confirmed disease progression assessed by investigator.
  Arms: cCRT plus placebo followed by durvalumab
Drug: Etoposide — Participants received etoposide 50 mg/m^2 intravenously over a minimum of 30 minutes up to 60 minutes daily on Day 1 to 5 and Day 29 to 33 during cCRT.
Drug: Pemetrexed — Participants received pemetrexed at a dose of 500 mg/m^2 intravenously over 10 minutes or according to local standards on Days 1, 22, and 43 during cCRT.
Drug: Carboplatin — Participants received carboplatin intravenously based on area under curve (AUC) 2 over 30 minutes on Day 1, Day 8, Day 15, Day 22, Day 29, Day 36, and Day 43 during cCRT.
Drug: Paclitaxel — Participants received paclitaxel intravenously at a dose of 45 mg/m^2 over 60 minutes on Day 1, Day 8, Day 15, Day 22, Day 29, Day 36, and Day 43 during cCRT.
Drug: Cisplatin — In combination with etoposide, participants received cisplatin 50 mg/m^2 intravenously over 60 minutes on Days 1, 8, 29, and 36 during cCRT. In combination with pemetrexed, participants received cisplatin 75 mg/m2 intravenously over 60 minutes on Days 1, 22, and 43 during cCRT.
Radiation: Intensity Modulated Radiation Therapy (IMRT) — Participants received IMRT 5 fractions per week for about 6 weeks (Total 60 gray [Gy]).

SUMMARY:
The main purpose of this study was to evaluate safety and efficacy in participants treated with concomitant chemoradiation therapy (cCRT) plus M7824 followed by M7824 compared to cCRT plus placebo followed by durvalumab.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically documented NSCLC who present with Stage III locally advanced, unresectable disease (International Association for the Study of Lung Cancer Staging Manual in Thoracic Oncology
* Participants with tumor harboring an Epidermal growth factor receptor (EGFR) sensitizing (activating) mutation, Anaplastic lymphoma kinase (ALK) translocation, ROS-1 rearrangement are eligible.
* Participants must have adequate pulmonary function defined as a forced expiratory volume in 1 second (FEV1) greater than equals to (>=) 1.2 liters or >= 50% of predicted normal volume measured within 3 weeks prior to randomization.
* Adequate hematological, hepatic and renal function as defined in the protocol
* Contraceptive use by males or females will be consistent with local regulations on contraception methods for those participating in clinical studies

Exclusion Criteria:

* Participants with Mixed small cell with non-small cell lung cancer histology
* Recent major surgery within 4 weeks prior to entry into the study
* Significant acute or chronic infections including human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome, Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection and active tuberculosis
* Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization
* Active autoimmune disease that has required systemic treatment in past 1 year (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs)
* Any prior systemic cytotoxic chemotherapy for their NSCLC or any antibody or drug targeting T-cell coregulatory proteins

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2023-02-17 (Actual); Study Completion 2023-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (104):
- United States (21):
  - University of California Irvine Medical Center, Orange, California
  - UCLA Hematology Oncology - Main Site - 2020 Santa Monica, Santa Monica, California
  - University of Colorado Health - Memorial Hospital - Memorial Hospital, Colorado Springs, Colorado
  - Hematology Oncology Associates, Fort Collins, Colorado
  - Lynn Cancer Institute Center, Boca Raton, Florida
  - Holy Cross Hospital - Michael and Dianne Bienes CCC, Fort Lauderdale, Florida
  - Sylvester Comprehensive Cancer Center - University of Miami Health System, Miami, Florida
  - The University of Chicago Medical Center, Chicago, Illinois
  - American Health Network of Indiana, LLC, Indianapolis, Indiana
  - Franciscan St. Francis Health Cancer Center, Indianapolis, Indiana
  - Baptist Health Lexington Oncology Associates, Lexington, Kentucky
  - University of Maryland - DUPLICATE/Pediatric Surgery, Baltimore, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Columbia University Medical Center, New York, New York
  - Hematology Oncology Center of Nyack Hospital, Nyack, New York
  - FirstHealth of the Carolinas, Inc., Pinehurst, North Carolina
  - The James Cancer Hospital and Solove Research Institute, Columbus, Ohio
  - UPMC Cancer Center, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center - Unit 432 Thoracic Head and Neck Medical Oncology, Houston, Texas
- Argentina (2):
  - Sanatorio Allende, Córdoba
  - Centro Polivalente de Asistencia e Inv. Clinica CER, San Juan
- Australia (11):
  - Bendigo Hospital, Bendigo
  - The Townsville Hospital, Douglas
  - Calvary Central Districts Hospital, Elizabeth Vale
  - St Vincent's Hospital Melbourne - PARENT, Fitzroy
  - University Hospital Geelong - PARENT, Geelong
  - Austin Health, Heidelberg Heights
  - Centro de Investigacion Pergamino SA, Pergamino
  - Prince of Wales Hospital, Randwick
  - Sunshine Hospital, St Albans
  - Royal North Shore Hospital, St Leonards
  - South West Healthcare - South West Oncology, Warrnambool
- Belgium (4):
  - UZ Leuven, Leuven
  - Clinique et Maternite St Elisabeth Namur, Namur
  - AZ Delta, Roeselare
  - CHU Mont-Godinne, Yvoir
- Brazil (7):
  - Hospital de Câncer de Barretos - Fundação Pio XII, Barretos
  - Clínica de Neoplasias Litoral Ltda., Itajaí
  - HGB - Hospital Giovanni Battista - Mãe de Deus Center - Centro de Pesquisa Clínica - Instituto do Câncer, Porto Alegre
  - Hospital São Lucas da PUCRS, Porto Alegre
  - COI - Clínicas Oncológicas Integradas, Rio de Janeiro
  - A. C. Camargo Cancer Center - Fundação Antônio Prudente, São Paulo
  - ICESP - Instituto do Câncer do Estado de São Paulo Octavio Frias de Oliveira, São Paulo
- BC Cancer Agency Center for the Southern Interior, Kelowna, Canada
- China (3):
  - Peking University Cancer Hospital, Beijing
  - Jilin Cancer Hospital - Oncology, Changchun
  - Hangzhou First People's Hospital, Hangzhou
- Fakultni nemocnice Olomouc - Dept of Onkologicka klinika, Olomouc, Czechia
- France (4):
  - Centre Hospitalier de la Côte Basque - Service de Pneumologie, Bayonne
  - Hôpital Nord - AP-HM Marseille# - Service d'Oncologie Multidisciplinaire, Marseille
  - Institut Curie - Centre de Lutte Contre le Cancer (CLCC) de Paris - Service d'Oncologie Médicale, Paris
  - CHU Nantes - Hôpital Guillaume et René Laënnec - Service de Pneumologie, Saint-Herblain
- Germany (2):
  - Asklepios Klinik Harburg - Medizinische Abteilung I, Hamburg
  - Pius-Hospital Oldenburg - Klinik f. Haematologie und Onkologie, Oldenburg
- Japan (12):
  - Nippon Medical School Hospital - Dept of Respiratory Medicine, Bunkyō City
  - Tokyo Metropolitan Cancer and Infectious diseases Center Komagome Hospital - Dept of Respiratory Medicine, Bunkyō City
  - Saitama Medical University International Medical Center - Dept of Respiratory Medicine, Hidaka-shi
  - National Cancer Center Hospital East - Dept of Respiratory Medicine, Kashiwa-shi
  - Kobe City Hospital Organization Kobe City Medical Center General Hospital - Dept of Respiratory Medicine, Kobe
  - Cancer Institute Hospital of JFCR - Dept of Respiratory Medicine, Kōtoku
  - Kurume University Hospital - Dept of Lung Cancer Center, Kurume-shi
  - Aichi Cancer Center Hospital - Dept of Respiratory Medicine, Nagoya
  - Osaka Medical Center for Cancer and Cardiovascular Diseases, Osaka
  - Kindai University Hospital (13859), Osakasayama-shi
  - Shizuoka Cancer Center, Sunto-gun
  - Kanagawa Cancer Center - Dept of Respiratory Medicine, Yokohama
- Netherlands (8):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Meander Medisch Centrum - Dep of Pulmonology, Amersfoort
  - Amphia Ziekenhuis - PARENT - Parent, Breda
  - Martini ziekenhuis, Groningen
  - Ziekenhuis St. Jansdal, Harderwijk
  - St. Antonius Ziekenhuis - Dept Pulmonology - Nieuwegein, Nieuwegein
  - St. Elisabeth Ziekenhuis - Parent, Tilburg
  - ISALA Klinieken Locatie Sophia, Zwolle
- South Korea (6):
  - Keimyung University Dongsan Hospital, Daegu
  - Seoul National University Bundang Hospital, Seongnam
  - Asan Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Severance Hospital, Yonsei University, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
- Spain (18):
  - Hospital del Mar - Servicio de Oncologia, Barcelona
  - Hospital Universitari Quiron Dexeus - Servicio de Oncologia Medica, Barcelona
  - Hospital Universitari Vall d'Hebron - Dept of Oncology, Barcelona
  - ICO l´Hospitalet - Hospital Duran i Reynals - Servicio de Oncologia, L'Hospitalet de Llobregat
  - Clinica Universidad de Navarra (MAD) - Oncology Service, Madrid
  - Hospital Universitario 12 de Octubre - Servicio de Oncologia, Madrid
  - Hospital Universitario Clinico San Carlos - Servicio de Oncologia, Madrid
  - Hospital Universitario HM Madrid Sanchinarro - Servicio de Oncologia, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda
  - Hospital Regional Universitario de Malaga, Málaga
  - Clinica Universidad de Navarra, Pamplona
  - Complejo Hospitalario Universitario de Santiago - Servicio de Oncologia Medica, Santiago de Compostela
  - Hospital Universitario Nuestra Señora de Valme - Servicio de Oncologia, Seville
  - Hospital Universitario Virgen del Rocio - Servicio de Oncologia, Seville
  - Hospital Universitario Virgen Macarena - Servicio de Oncologia, Seville
  - Hospital Clinico Universitario de Valencia - Servicio de Hematologia y Oncologia Medica, Valencia
  - Hospital Universitari i Politecnic La Fe - Servicio de Oncologia Medica, Valencia
  - Hospital Alvaro Cunqueiro - Servicio de Oncologia, Vigo
- Taiwan (4):
  - Taichung Veterans General Hospital, Taichung
  - Chi Mei Medical Center, Liou Ying, Tainan
  - National Taiwan University Hospital, Taipei
  - Tri-Service General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Within six months after the approval of a new product or a new indication for an approved product in both the United States and the European Union
Access Criteria: Qualified scientific and medical researchers can request the data. Such requests must be submitted in writing to the company's portal and will be internally reviewed regarding criteria for researchers' qualification and legitimacy of the research proposal.
URL: http://bit.ly/IPD21

REFERENCES:
- [Derived] Huang Y, Zhao JJ, Soon YY, Wong A, Aminkeng F, Ang Y, Asokumaran Y, Low JL, Lee M, Choo JRE, Chan G, Kee A, Tay SH, Goh BC, Soo RA. Real-world experience of consolidation durvalumab after concurrent chemoradiotherapy in stage III non-small cell lung cancer. Thorac Cancer. 2022 Nov;13(22):3152-3161. doi: 10.1111/1759-7714.14667. Epub 2022 Sep 30. PMID 36177913
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200647_0005
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First participant signed informed consent: 16-Apr-2019, Clinical data cut-off: 21-Jul-2021.
Groups:
- cCRT Plus M7824 Followed by M7824: Participants received Concomitant Chemoradiotherapy (cCRT): Cisplatin/Etoposide (50 milligrams per square meter (mg/m^2) of Cisplatin intravenously over 60 minutes on Days 1, 8, 29, and 36 with 50 mg/m^2 intravenously of Etoposide over a minimum of 30 minutes up to 60 minutes daily on Day 1 to 5 and Day 29 to 33 during cCRT or Carboplatin/Paclitaxel (carboplatin intravenously based on area under curve (AUC) 2 over 30 minutes on Day 1, Day 8, Day 15, Day 22, Day 29, Day 36, and Day 43 with 45 mg/m^2 of Paclitaxel over 60 minutes on Day 1, Day 8, Day 15, Day 22, Day 29, Day 36, and Day 43 during cCRT or Cisplatin/Pemetrexed (50 mg/m^2 of Cisplatin intravenously over 60 minutes on Days 1, 8, 29, and 36 with 500 mg/m^2 of Pemetrexed intravenously over 10 minutes or according to local standards on Days 1, 22, and 43 during cCRT concomitant with Intensity Modulated Radiation Therapy 5 (IMRT 5), fractions per week for about 6 weeks (Total 60 gray [Gy]) in combination with intravenous infusion of 1200 mg of M7824 over 1 hour every 2 weeks (q2w) during cCRT and up to 1 year after cCRT until unacceptable toxicity, confirmed disease progression assessed by investigator.
- cCRT Plus Placebo Followed by Durvalumab: Participants received Concomitant Chemoradiotherapy (cCRT): Cisplatin/Etoposide (50 mg/m^2) of Cisplatin intravenously over 60 minutes on Days 1, 8, 29, and 36 with 50 mg/m^2 intravenously of Etoposide over a minimum of 30 minutes up to 60 minutes daily on Day 1 to 5 and Day 29 to 33 during cCRT or Carboplatin/Paclitaxel, carboplatin intravenously based on area under curve (AUC) 2 over 30 minutes on Day 1, Day 8, Day 15, Day 22, Day 29, Day 36, and Day 43 with 45 mg/m^2 of Paclitaxel over 60 minutes on Day 1, Day 8, Day 15, Day 22, Day 29, Day 36, and Day 43 during cCRT or Cisplatin/Pemetrexed, 50 mg/m^2 of Cisplatin intravenously over 60 minutes on Days 1, 8, 29, and 36 with 500 mg/m^2 of Pemetrexed intravenously over 10 minutes or according to local standards on Days 1, 22, and 43 during cCRT concomitant with Intensity Modulated Radiation Therapy 5 (IMRT 5), fractions per week for about 6 weeks (Total 60 gray [Gy]) in combination with intravenous infusion of placebo matched to M7824 over 1 hour q2w during cCRT followed by intravenous infusion of durvalumab 10 milligram per kilogram (mg/Kg) over 1 hour q2w up to 1 year after cCRT until unacceptable toxicity, confirmed disease progression assessed by investigator.
Period: Overall Study
Arm/Group | cCRT Plus M7824 Followed by M7824 | cCRT Plus Placebo Followed by Durvalumab
Started | 75 | 78
Treated | 74 | 77
Completed | 74 | 77
Not Completed | 1 | 1
Not completed — Randomized but not treated | 1 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all participants who were randomized to study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | cCRT Plus M7824 Followed by M7824 | cCRT Plus Placebo Followed by Durvalumab | Total
Number analyzed (Participants) | 75 | 78 | 153
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.7 (9.35) | 64.9 (8.94) | 64.8 (9.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 16 | 36
  Male | 55 | 62 | 117
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 8
  Not Hispanic or Latino | 70 | 74 | 144
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 25 | 34 | 59
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 48 | 41 | 89
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) According to Response Evaluation Criteria in Solid Tumors (RECIST Version 1.1) Assessed by Investigator
Description: PFS was defined as the time from randomization to the date of first documentation of disease progression (PD) or death due to any cause, whichever occurred first. PD: At least a 20 percent (%) increase in the sum of the longest diameter (SLD) taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions. PFS was analyzed by using the Kaplan-Meier method.
Time Frame: Time from randomization to the date of first documentation of PD or death, assessed approximately up to 27 months
Population: Full Analysis Set (FAS) included all participants who were randomized to study treatment.
Measure: Median (Full Range); unit: months
Arm/Group | cCRT Plus M7824 Followed by M7824 | cCRT Plus Placebo Followed by Durvalumab
Number analyzed (Participants) | 75 | 78
months | 3.7 [1.9 to 5.6] | 3.7 [1.8 to 3.9]

2. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Related Adverse Events
Description: Adverse Event (AE) was defined any untoward medical occurrence in a participant administered with a study drug, which does not necessarily have a causal relationship with this treatment. Serious AE was defined AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial/prolonged inpatient hospitalization; congenital anomaly/birth defect. TEAEs: TEAEs was defined as events with onset date or worsening during the on-treatment period. TEAEs included serious AEs and non-serious AEs. Treatment-related TEAEs: reasonably related to the study intervention.
Time Frame: Time from randomization up to data cut off (assessed up to 27 months)
Population: Safety (SAF) Analysis Set included all participants who were administered any dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | cCRT Plus M7824 Followed by M7824 | cCRT Plus Placebo Followed by Durvalumab
Number analyzed (Participants) | 74 | 77
Participants
  Participants with TEAEs | 70 | 74
  Participants with immunotherapy related TEAE | 48 | 48
  Participants with cisplatin/etoposide chemotherapy regimen related TEAE | 7 | 11
  Participants with carboplatin/paclitaxel chemotherapy regimen related TEAE | 46 | 47
  Participants with cisplatin/pemetrexed chemotherapy regimen related TEAE | 15 | 11
  Participants with radiotherapy related TEAE | 59 | 60

3. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival was defined as the time from randomization to the date of death due to any cause. The overall survival was analyzed by using the Kaplan-Meier method.
Time Frame: Time from randomization to the date of death due to any cause, assessed up to 27 months
Population: FAS included all participants who were randomized to study treatment.
Measure: Median (Full Range); unit: months
Arm/Group | cCRT Plus M7824 Followed by M7824 | cCRT Plus Placebo Followed by Durvalumab
Number analyzed (Participants) | 75 | 78
months | 4.6 [0.1 to 22.3] | 4.3 [0.3 to 22.7]

4. Secondary Outcome: Objective Response Rate (ORR) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as Assessed by Investigator
Description: ORR was defined as the percentage of participants who had achieved complete response (CR) or partial response (PR) as the best overall response according to RECIST v1.1as adjudicated by the Investigator. CR: Complete Response (CR) defined as disappearance of all target and non-target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. Partial response (PR) defined as at least a 30% decrease in the sum of diameters of target lesions.
Time Frame: Time from randomization up to data cut off (assessed up to 27 months)
Population: FAS included all participants who were randomized to study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | cCRT Plus M7824 Followed by M7824 | cCRT Plus Placebo Followed by Durvalumab
Number analyzed (Participants) | 75 | 78
percentage of participants | 29.3 [19.4 to 41.0] | 32.1 [21.9 to 43.6]

5. Secondary Outcome: Duration of Response (DOR) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as Assessed by Investigator
Description: DOR was defined as the time from first documentation of objective response (Complete Response [CR] or Partial Response [PR]) to the date of first documentation of progression disease (PD) or death due to any cause, whichever occurred first. CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the SLD of all lesions. PD: At least a 20 percent (%) increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions. DOR was determined according to RECIST v1.1 and assessed by IRC. Results were calculated based on Kaplan-Meier estimates.
Time Frame: Time from first documentation of objective response to the date of first documentation of PD or death due to any cause, assessed approximately up to 27 months
Population: Due to early termination of the study, the data for this outcome measure was not collected.
Arm/Group | cCRT Plus M7824 Followed by M7824 | cCRT Plus Placebo Followed by Durvalumab
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Immediate Observed Serum Concentration at End of Infusion (Ceoi) of M7824
Description: Ceoi is the serum concentration observed immediately at the end of infusion. This was taken directly from the observed M7824 concentration-time data.
Time Frame: Pre-dose, 30 minutes after end of infusion on Day 1, 15, 29, 57, 85, 127, 157, 343
Population: Based on recommendations by an external Independent Data Monitoring Committee (IDMC), Sponsor decided to discontinue this clinical study. Subsequently, the data for this outcome measure was not collected and analyzed.
Arm/Group | cCRT Plus M7824 Followed by M7824 | cCRT Plus Placebo Followed by Durvalumab
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Serum Concentration Immediately Before Next Dosing (Ctrough) of M7824
Description: Ctrough was the serum concentration observed immediately before next dosing.
Time Frame: Pre-dose, 30 minutes after end of infusion on Day 1, 15, 29, 57, 85, 127, 157, 343
Population: as for outcome 6
Arm/Group | cCRT Plus M7824 Followed by M7824 | cCRT Plus Placebo Followed by Durvalumab
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Number of Participants With Positive Antidrug Antibodies (ADA)
Description: Serum samples were analyzed by a validated assay method to detect the presence of antidrug antibodies (ADA). Number of participants with positive ADA were reported.
Time Frame: Time from randomization up to data cut off (assessed up to 27 months)
Population: as for outcome 6
Arm/Group | cCRT Plus M7824 Followed by M7824 | cCRT Plus Placebo Followed by Durvalumab
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Time from randomization up to data cut off (assessed up to 27 months)
Description: Safety (SAF) Analysis Set included all participants who were administered any dose of any study intervention. All-Cause Mortality was assessed on Full Analysis Set, Serious Adverse Events or Other (Not Including Serious) Adverse Events was done on Safety (SAF) Analysis Set.
Arm/Group | cCRT Plus M7824 Followed by M7824 | cCRT Plus Placebo Followed by Durvalumab
All-Cause Mortality (participants affected / at risk) | 13/75 | 5/78
Serious Adverse Events (participants affected / at risk) | 43/74 | 31/77
Other Adverse Events (participants affected / at risk) | 68/74 | 72/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | cCRT Plus M7824 Followed by M7824 (N=74) | cCRT Plus Placebo Followed by Durvalumab (N=77)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Myelosuppression (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal vascular malformation haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 3 (6)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (6) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0)
Disease progression (General disorders) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 1 (2) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 2 (3)
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Contrast media allergy (Immune system disorders) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (2) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 3 (5) | 4 (4)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 1 (1)
Septic shock (Infections and infestations) | 2 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radiation mucositis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radiation oesophagitis (Injury, poisoning and procedural complications) | 3 (7) | 2 (2)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Glomerular filtration rate decreased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain stem haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 1 (1)
Thoracic outlet syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 (8) | 6 (9)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | cCRT Plus M7824 Followed by M7824 (N=74) | cCRT Plus Placebo Followed by Durvalumab (N=77)
Anaemia (Blood and lymphatic system disorders) | 38 (49) | 32 (53)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 9 (13) | 10 (12)
Lymphopenia (Blood and lymphatic system disorders) | 4 (4) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 20 (27) | 15 (18)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 11 (16) | 7 (8)
Angina pectoris (Cardiac disorders) | 2 (3) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 4 (4) | 7 (7)
Hypopituitarism (Endocrine disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 2 (2) | 6 (6)
Thyroiditis (Endocrine disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 0 (0)
Abdominal rigidity (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 3 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 23 (26) | 34 (43)
Dental caries (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 12 (14) | 12 (13)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 5 (5) | 4 (4)
Dysphagia (Gastrointestinal disorders) | 9 (10) | 5 (5)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 3 (3) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 5 (5)
Gingival bleeding (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 26 (29) | 29 (35)
Odynophagia (Gastrointestinal disorders) | 5 (6) | 6 (7)
Oesophageal ulcer (Gastrointestinal disorders) | 2 (2) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 15 (15) | 24 (25)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 3 (3) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 9 (9) | 3 (3)
Vomiting (Gastrointestinal disorders) | 9 (12) | 6 (7)
Asthenia (General disorders) | 13 (19) | 6 (6)
Catheter site pruritus (General disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 2 (2) | 0 (0)
Chills (General disorders) | 1 (1) | 4 (4)
Fatigue (General disorders) | 5 (5) | 14 (15)
Feeling hot (General disorders) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Generalised oedema (General disorders) | 1 (1) | 1 (1)
Hyperthermia (General disorders) | 1 (1) | 0 (0)
Infusion site extravasation (General disorders) | 1 (1) | 0 (0)
Infusion site reaction (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 5 (6) | 6 (6)
Mucosal haemorrhage (General disorders) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 5 (6) | 2 (3)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 18 (22) | 10 (11)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (2)
Cytomegalovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 2 (2) | 0 (0)
Empyema (Infections and infestations) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 2 (4) | 0 (0)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 2 (2) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Molluscum contagiosum (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 1 (2) | 0 (0)
Oesophageal infection (Infections and infestations) | 1 (1) | 0 (0)
Onychomycosis (Infections and infestations) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1) | 1 (1)
Oral fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Peri-implantitis (Infections and infestations) | 1 (1) | 0 (0)
Periodontitis (Infections and infestations) | 1 (1) | 1 (1)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 8 (9) | 3 (3)
Post-acute COVID-19 syndrome (Infections and infestations) | 0 (0) | 1 (1)
Pseudomembranous colitis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2)
Tinea infection (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 6 (10) | 3 (3)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radiation fibrosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radiation fibrosis - lung (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Radiation mucositis (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Radiation oesophagitis (Injury, poisoning and procedural complications) | 13 (13) | 13 (15)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 7 (7) | 9 (12)
Radiation skin injury (Injury, poisoning and procedural complications) | 5 (5) | 10 (10)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 6 (10) | 9 (11)
Alpha hydroxybutyrate dehydrogenase increased (Investigations) | 1 (1) | 0 (0)
Amylase increased (Investigations) | 5 (11) | 1 (3)
Anti-transglutaminase antibody increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 6 (7) | 7 (11)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 2 (3)
Blood bilirubin increased (Investigations) | 3 (4) | 3 (5)
Blood cholesterol increased (Investigations) | 1 (1) | 4 (4)
Blood creatine increased (Investigations) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 4 (8) | 2 (2)
Blood creatinine increased (Investigations) | 4 (4) | 3 (4)
Blood glucose increased (Investigations) | 2 (3) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (2) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1) | 1 (1)
Blood triglycerides increased (Investigations) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 2 (5) | 5 (9)
Brain natriuretic peptide increased (Investigations) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 1 (2) | 2 (2)
Fibrin D dimer increased (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 5 (7) | 7 (13)
Gastric pH decreased (Investigations) | 0 (0) | 1 (1)
Glomerular filtration rate decreased (Investigations) | 1 (2) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 8 (9) | 1 (1)
Lung diffusion test decreased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 11 (16) | 13 (23)
Neutrophil count decreased (Investigations) | 17 (28) | 20 (36)
Platelet count decreased (Investigations) | 11 (16) | 13 (21)
Procalcitonin increased (Investigations) | 1 (1) | 0 (0)
Protein total decreased (Investigations) | 0 (0) | 1 (1)
Prothrombin time prolonged (Investigations) | 1 (2) | 0 (0)
Pulmonary function test decreased (Investigations) | 1 (1) | 2 (2)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 1 (1)
Total bile acids increased (Investigations) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 8 (9) | 8 (8)
Weight increased (Investigations) | 0 (0) | 2 (2)
White blood cell count decreased (Investigations) | 24 (37) | 29 (59)
White blood cell count increased (Investigations) | 1 (1) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 17 (20) | 16 (17)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 6 (7) | 5 (7)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 4 (7)
Hyperuricaemia (Metabolism and nutrition disorders) | 3 (4) | 3 (6)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 10 (16) | 5 (6)
Hypocalcaemia (Metabolism and nutrition disorders) | 4 (4) | 2 (3)
Hypochloraemia (Metabolism and nutrition disorders) | 1 (1) | 4 (6)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4) | 3 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 (5) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 6 (13) | 9 (15)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 5 (5) | 0 (0)
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 3 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 4 (4)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (5) | 0 (0)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral microhaemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 5 (5)
Dizziness exertional (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 4 (5)
Neuropathy peripheral (Nervous system disorders) | 2 (2) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 2 (2)
Tremor (Nervous system disorders) | 2 (2) | 0 (0)
Device malfunction (Product Issues) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Anxiety disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 9 (10) | 9 (11)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (2)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Erection increased (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 14 (16)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 7 (7)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 13 (16) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 3 (3)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 6 (9) | 6 (6)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 10 (12)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 2 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (6) | 7 (7)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 5 (7) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Neurodermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 13 (18) | 8 (8)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 19 (25) | 6 (7)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
Skin reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin toxicity (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 2 (2)
Hypotension (Vascular disorders) | 4 (4) | 4 (5)
Intermittent claudication (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 2 (2) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1)
Phlebitis superficial (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-06-22): https://cdn.clinicaltrials.gov/large-docs/02/NCT03840902/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-22): https://cdn.clinicaltrials.gov/large-docs/02/NCT03840902/SAP_001.pdf